CLINICAL TRIAL: NCT01104740
Title: Dengue Seroprevalence Study in Blood Donors in the French West Indies
Acronym: DengSeroprevAn
Status: Completed | Type: Observational
Sponsor: Etablissement Français du Sang, Martinique (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Clinique Antilles-Guyane (Other)
Responsible Party: Principal Investigator, RICHARD, Directrice EFS Martinique, Etablissement Français du Sang, Martinique
Other Study IDs: 10/B/01; 2010-A00385-34 (Other: AFSSAPS (ANSM))
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Blood Donors; Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Biological sample collection — Blood (serum) sample collection

SUMMARY:
Dengue is an infectious disease most prevalent in the world. This disease is endemic in the Caribbean, with an increase in seasonal rains. Several outbreaks have been observed in recent years, in 2001, 2005 and 2007, during which further particularly virulent serotypes have emerged. The clinical expression of dengue fever is variable, ranging from no symptoms to a classical form with fever, and even of severe or lethal bleeding. With the possible existence of silent forms of the disease, there are no data identifying the current level of protection of the population in Martinique / Guadeloupe.

DETAILED DESCRIPTION:
1. Principal objective:

   To estimate the prevalence of the specific antibodies of the dengue (IgG) in blood donors in the French West Indies.
2. Secondary objective:

To specify the serotypic specificity of the anti-dengue antibodies detected during the study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for blood donation following the French legislation,
* Resident in Martinique /Guadeloupe for at least one year
* Consent signed

Exclusion Criteria:

* Not Eligible for blood donation following the French legislation,
* Not Resident in Martinique / Guadeloupe for at least one year
* Consent not signed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult, résidents in Martinique/ Guadeloupe (french west indies), aged 18 to 65 years coming to give their blood in one of the building or mobile collection facilities of the French Blood Establishment in French West Indies.
Sampling Method: Non-Probability Sample
Enrollment: 817 (Actual)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Presence or not of dengue virus-specific immunoglobulin G antibodies | 1 day

SECONDARY OUTCOMES:
Characterization of dengue virus serotype-specific IgG | 1 day
  Characterization of dengue virus serotype-psecific IgG whendengue virus serotype-specific immunoglobulin G antibodies Test is positive

CONTACTS AND LOCATIONS:
Overall Officials: Pascale RICHARD, MD, Principal Investigator — French Blood Establishment of Martinique
Locations (2):
- French Blood Establishment of Guadeloupe, Pointe-à-Pitre, Guadeloupe
- French Blood Establishment of Martinique, Fort-de-France, Martinique